CLINICAL TRIAL: NCT05905939
Title: A Multicenter Observational Retrospective Study of Therapeutic Approaches and Clinical Outcomes in Real Clinical Practice in Russian Patients With Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Metastatic Breast Cancer
Brief Title: HER2(Human Epidermal Growth Factor Receptor 2) -Positive Metastatic Breast Cancer in Russia
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133HR00027
Record Dates: First submitted 2023-06-01; First posted 2023-06-15 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

SUMMARY:
Planned study population consists of approximately 1,000 adult patients with HER2-positive mBC receiving anti-HER2 therapy in about 50 oncological centers (in each center it is expected to recruit about 20 patients) in different regions in order to provide representative study sample. Patients will be included consecutively from the least recent diagnosis (within defined time period).

Planned retrospective follow-up period for 1 patient is a period starting from the date of mBC diagnosis until end study or until patient's death, whichever occurs first. End of study will be at least 12 months after the latest date of mBC diagnosis to ensure all patients have the opportunity to contribute at least 12 months of data.

DETAILED DESCRIPTION:
Planned study population consists of approximately 1,000 adult patients with HER2-positive mBC receiving anti-HER2 therapy in about 50 oncological centers (in each center it is expected to recruit about 20 patients) in different regions in order to provide representative study sample. Patients will be included consecutively from the least recent diagnosis (within defined time period).

Planned retrospective follow-up period for 1 patient is a period starting from the date of mBC diagnosis until end study or until patient's death, whichever occurs first. End of study will be at least 12 months after the latest date of mBC diagnosis to ensure all patients have the opportunity to contribute at least 12 months of data.

Only patients who were diagnosed between the 1st July 2021 and 1st July 2022 will be included. Patients should have at least 12 months of follow-up data. In case patient died within the first 12 months of diagnosis, these data from date of mBC diagnosis until patient's death should also be included. It will be multicenter study

ELIGIBILITY:
Inclusion Criteria:

* Patients with HER2-positive mBC who are receiving or have started any anti-HER2 therapy (except for trastuzumab deruxtecan) at the time of inclusion;
* The diagnosis of mBC was established between the 1st July 2021 and the 1st July 2022;
* Patients with the availability of at least 12 months of follow-up data (from the index data) in the medical records at the participating site, unless patient died within the first 12 months of diagnosis;
* Age ≥ 18 years at the time of inclusion.

Exclusion Criteria:

* Presence of other malignancies within period since diagnosis until the timepoint of data collection;
* Patients receiving trastuzumab deruxtecan currently or in the anamnesis;
* The participation in any randomized controlled trial within period since diagnosis until end of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This non-interventional multicenter observational study will include 1,000 adult patients with HER2-positive mBC receiving anti-HER2 therapy (except for trastuzumab deruxtecan).
  Patients will be included in about 50 oncological centers (in each center it is expected to recruit about 20 patients) in various regions of Russian Federation
Sampling Method: Non-Probability Sample
Enrollment: 774 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
To describe the clinical and demographic profiles of patients with HER2-positive mBC receiving anti-HER2 therapy (except for trastuzumab deruxtecan) in the Russian Federation | up to 6 month
  Demographics characteristics : age(years)
To describe the clinical and demographic profiles of patients with HER2-positive mBC receiving anti-HER2 therapy (except for trastuzumab deruxtecan) in the Russian Federation | up to 6 month
  - Demographics characteristics : gender
To describe the clinical and demographic profiles of patients with HER2-positive mBC receiving anti-HER2 therapy (except for trastuzumab deruxtecan) in the Russian Federation | up to 6 month
  - Demographics characteristics : body mass index [BMI]);
To describe the clinical and demographic profiles of patients with HER2-positive mBC receiving anti-HER2 therapy (except for trastuzumab deruxtecan) in the Russian Federation | up to 6 month
  Clinical characteristics, including BC history, family and personal oncology history
To describe the clinical and demographic profiles of patients with HER2-positive mBC receiving anti-HER2 therapy (except for trastuzumab deruxtecan) in the Russian Federation | up to 6 month
  Clinical characteristics: ECOG status
To describe the clinical and demographic profiles of patients with HER2-positive mBC receiving anti-HER2 therapy (except for trastuzumab deruxtecan) in the Russian Federation | up to 6 month
  Clinical characteristics: HER2, estrogen receptor (ER), progesterone receptor (PR) expression status, Ki67 expression status (in %)
To describe the clinical and demographic profiles of patients with HER2-positive mBC receiving anti-HER2 therapy (except for trastuzumab deruxtecan) in the Russian Federation | up to 6 month
  Clinical characteristics: number of metastatic sites and localization

SECONDARY OUTCOMES:
To describe data on the diagnostic algorithms and therapeutic tactics in patients with HER2-positive mBC in routine practice in the Russian Federation | up to 6 month
  - Proportion of patients with different diagnostic method(s) used for the diagnosis;
To describe data on the treatment approach in patients with HER2-positive mBC in routine practice in the Russian Federation | up to 6 month
  * Anticancer therapy;
  * Concomitant therapy.
To assess the treatment outcomes of patients with HER2-positive mBC in routine practice in the Russian Federation | up to 6 month
  -Number of therapy lines, schemes and duration;
To describe data on the diagnostic algorithms and therapeutic tactics in patients with HER2-positive mBC in routine practice in the Russian Federation | up to 6 month
  - Proportion of patients treated for early BC (if conducted).
To assess the treatment outcomes of patients with HER2-positive mBC in routine practice in the Russian Federation | up to 6 month
  -Reasons for anticancer therapy discontinuation, if applicable;
To assess the treatment outcomes of patients with HER2-positive mBC in routine practice in the Russian Federation | up to 6 month
  -Time to treatment discontinuation (TTD), defined as the median time from the starting first line therapy to the treatment discontinuation from any cause;

CONTACTS AND LOCATIONS:
Locations (29):
- Russia (29):
  - Research Site, Arkhangelsk
  - Research Site, Barnaul
  - Research Site, Belgorod
  - Research Site, Chelyabinsk
  - Research Site, Grozny
  - Research Site, Irkutsk
  - Research Site, Kaluga
  - Research Site, Kchabarovsk
  - Research Site, Khanty-Mansiysk
  - Research Site, Kommunarka
  - Research Site, Kostroma
  - Research Site, Krasnodar
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Perm
  - Research Site, Pyatigorsk
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Sakhalin
  - Research Site, Saransk
  - Research Site, Sochi
  - Research Site, Surgut
  - Research Site, Tomsk
  - Research Site, Tver'
  - Research Site, Ufa
  - Research Site, Ulan-Ude
  - Research Site, Vladivostok
  - Research Site, Volgograd
  - Research Site, Yaroslavl

REFERENCES:
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D133HR00027&attachmentIdentifier=b6ce4fbd-054f-4442-994f-194cfa5edf36&fileName=D133HR00027_Study_report_synopsis_1.0_2025_03_24.pdf&versionIdentifier=